CLINICAL TRIAL: NCT04296474
Title: Follow up Study 5-6 Years After ILIT With 2 Concomitant Allergens, Birch and Grass
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lars Olaf Cardell (Other)
Responsible Party: Sponsor-Investigator, Lars Olaf Cardell, Professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Follow-up ILIT 2018/2645-32
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Serum Albumin, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active ILIT treated (Active Comparator): Patients that have received ILIT with birch and grass allergen 5-6 years previously
  Interventions: Drug: ALK Alutard 5-grasses and birch
- Non- AIT treated (Placebo Comparator): Patients that have received placebo ILIT 5-6 years previously and patients with birch and grass pollen induced allergic rhinitis that have not previously been treated with allergen immunotherapy (AIT).
  Interventions: Drug: ALK Diluent

INTERVENTIONS:
Drug: ALK Alutard 5-grasses and birch — Intralymphatic injections
  Other Names: Grass and birch allergen with aluminum adjuvant
  Arms: Active ILIT treated
Drug: ALK Diluent — intralymphatic injections
  Other Names: Human albumin
  Arms: Non- AIT treated

SUMMARY:
52 patients that had previously participated in the RDBPC study of intralymphatic immunotherapy (ILIT) with 2 concomitant allergens, birch and grass, with NCT02423707, were eligible for an open follow up 5-6 years after treatment.

DETAILED DESCRIPTION:
Bakground: Intralymphatic immunotherapy has been proposed as a new, more effective, modality for allergy immunotherapy. With ultrasound- guided injections into the lymph node the allergen is injected directly to the secondary lymphoid organ to stimulate the immune system. The protocol that has been used so far is three injections with one month interval. The effect have been evaluated in several studies with limited sample sized and the effect have been estimated to be in the same range as after conventinal subcutaneous immunotherapy. No long term follow up have been performed.

Objective: To investigate if the clinical improvement and immunological alterations is maintained 5-6 years after ILIT with two concomitant allergens, birch and grass.

Methods: 52 patients that had previously participated in the RDBPC study were asked to participate in this open follow up.

ELIGIBILITY:
Inclusion Criteria:

- Moderate to severe allergic rhinitis to birch and grass pollen defined with a positive skin prick test and elevated allergen specific IgE antibodies

Exclusion Criteria:

* uncontrolled or perennial asthma
* other pulmonary disease
* known autoimmune or collagen disease
* chronic infection
* other significant disease
* severe atopic dermatitis
* use of beta blockers or angiotensin converting enzyme inhibitors as antihypertensive medications
* symptomatic sensitization to house dust mite or furry animals with daily exposure
* chronic upper airways disease
* pregnancy
* nursing
* obesity with BMI >30
* withdrawn informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Nasal grass allergen provocation | 5-6 years after active or placebo ILIT
  The symptoms are recorded during 30 minutes after nasal spray with grass allergen

SECONDARY OUTCOMES:
Nasal birch allergen provocation | 5-6 years after active or placebo ILIT
  The symptoms are recorded during 30 minutes after nasal spray with grass allergen
Combined symptoms and medciations score | Pollen season 5-7 years after active or placebo ILIT
  Ranging from 0- no symptoms and medication, to 6- maximum symptoms and medication.
Rhinoconjunctivitis quality of life questionnaire | Pollen season 5-7 years after active or placebo ILIT
  Average score of 28 questions ranging from 0-no impairment of quality of life, to 6- maximum impairment of quality of life.
Sinonasal outcome test quality of life questionnaire | Pollen season 5-7 years after active or placebo ILIT
  Sum of 22 questions. The score ranges from 0-no impairment of quality of life, to 110- maximum impairment of quality of life.
Allergen specific IgE | 5-6 years after active or placebo ILIT
  Blood test
Allergen specific IgG4 | 5-6 years after active or placebo ILIT
  Blood test
T-cell and basophil activation | 5-6 years after active or placebo ILIT
  Blood samples and lymph node aspirates are investigated with flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Lars Olaf Cardell, Professor, Principal Investigator — Karolinska Institutet
Locations (3):
- Sweden (3):
  - Allergic Unit at the Department of Oto-Rhino-Laryngology at Skåne University Hospital Lund, Lund
  - Allergic Unit at the Department of Oto-Rhino-Laryngology at Skåne University Hospital Malmö, Malmo
  - ENT department, Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hellkvist L, Hjalmarsson E, Kumlien Georen S, Karlsson A, Lundkvist K, Winqvist O, Westin U, Cardell LO. Intralymphatic immunotherapy with 2 concomitant allergens, birch and grass: A randomized, double-blind, placebo-controlled trial. J Allergy Clin Immunol. 2018 Oct;142(4):1338-1341.e9. doi: 10.1016/j.jaci.2018.05.030. Epub 2018 Jun 13. No abstract available. PMID 29908212